CLINICAL TRIAL: NCT03061214
Title: Efficacy and Safety of Semaglutide Once-weekly Versus Sitagliptin Once-daily as add-on to Metformin in Subjects With Type 2 Diabetes. A 30-week Randomised, Double-blind, Double-dummy, Active-controlled, Parallel-group, Multi-centre and Multi-national Trial
Brief Title: Efficacy and Safety of Semaglutide Once-weekly Versus Sitagliptin Once-daily as add-on to Metformin in Subjects With Type 2 Diabetes (SUSTAIN - CHINA MRCT)
Acronym: SUSTAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-4114; U1111-1149-0432 (Other: World Health Organization (WHO)); CTR20161003 (Registry Identifier: China Drug Trials (China))
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Results first posted 2020-04-09 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Semaglutide 0.5 mg OW + sitagliptin placebo OD (Experimental)
  Interventions: Drug: Semaglutide 0.5 mg; Drug: Sitagliptin placebo
- Semaglutide 1 mg OW + sitagliptin placebo OD (Experimental)
  Interventions: Drug: Semaglutide 1.0 mg; Drug: Sitagliptin placebo
- Sitagliptin OD + semaglutide placebo 0.5 mg OW (Active Comparator)
  Interventions: Drug: Sitagliptin; Drug: Semaglutide placebo 0.5 mg
- Sitagliptin OD + semaglutide placebo 1 mg OW (Active Comparator)
  Interventions: Drug: Sitagliptin; Drug: Semaglutide placebo 1.0 mg

INTERVENTIONS:
Drug: Semaglutide 0.5 mg — Up to 0.5 mg semaglutide injected subcutaneously (s.c., under the skin) once-weekly (OW) for 30 weeks
  Arms: Semaglutide 0.5 mg OW + sitagliptin placebo OD
Drug: Semaglutide 1.0 mg — Up to 1.0 mg semaglutide injected subcutaneously once-weekly for 30 weeks
  Arms: Semaglutide 1 mg OW + sitagliptin placebo OD
Drug: Sitagliptin placebo — Sitagliptin placebo tablets taken once-daily for 30 weeks
  Arms: Semaglutide 0.5 mg OW + sitagliptin placebo OD; Semaglutide 1 mg OW + sitagliptin placebo OD
Drug: Sitagliptin — 100 mg sitagliptin tablets taken once-daily for 30 weeks
  Arms: Sitagliptin OD + semaglutide placebo 0.5 mg OW; Sitagliptin OD + semaglutide placebo 1 mg OW
Drug: Semaglutide placebo 0.5 mg — Semaglutide placebo (0.5 mg) injected subcutaneously once-weekly for 30 weeks
  Arms: Sitagliptin OD + semaglutide placebo 0.5 mg OW
Drug: Semaglutide placebo 1.0 mg — Semaglutide placebo (1.0 mg) injected subcutaneously once-weekly for 30 weeks
  Arms: Sitagliptin OD + semaglutide placebo 1 mg OW

SUMMARY:
This trial is conducted in Africa, Asia, Europe and South America. The aim of the trial is to compare the effect of once-weekly dosing of two dose levels of semaglutide versus sitagliptin 100 mg once-daily on glycaemic control after 30 weeks of treatment. Subjects will remain on their stable pre-trial metformin.

ELIGIBILITY:
Inclusion Criteria: - Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial - Male or female, age equal to or above 18 years at the time of signing informed consent - Subjects diagnosed with type 2 diabetes and on stable treatment in a period of 60 days prior to screening with metformin equal to or above 1500 mg (or maximum tolerated dose equal to or above 1000 mg). Stable is defined as unchanged medication and unchanged daily dose - HbA1c 7.0 - 10.5 % (53-91 mmol/mol) (both inclusive) Exclusion Criteria: - Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential not using an adequate contraceptive method throughout the trial including the 5 week follow-up period (adequate contraceptive measure as required by local regulation or practice) - Any disorder which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol - Treatment with glucose lowering agent(s) other than stated in the inclusion criteria in a period of 60 days before screening. An exception is short-term treatment (equal to or below 7 days in total) with insulin in connection with inter-current illness - History of chronic or idiopathic acute pancreatitis - Screening calcitonin value equal to or above 50 ng/L (pg/mL) - Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2) - Impaired renal function defined as estimated glomerular filtration rate (eGFR) below 60 ml/min/1.73 m^2 per modification of diet in renal disease (MDRD) formula (4 variable version) - Acute coronary or cerebrovascular event within 90 days before randomisation - Heart failure, New York Heart Association (NYHA) class IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 868 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- Brazil (3):
  - Novo Nordisk Investigational Site, Aparecida de Goiânia, Goiás
  - Novo Nordisk Investigational Site, Porto Alegre, Rio Grande do Sul
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
- China (27):
  - Novo Nordisk Investigational Site, Hefei, Anhui
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chongqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Fuzhou, Fujian
  - Novo Nordisk Investigational Site, Guangzhou, Guangdong
  - Novo Nordisk Investigational Site, Zhuhai, Guangdong
  - Novo Nordisk Investigational Site, Guiyang, Guizhou
  - Novo Nordisk Investigational Site, Qiqihar, Heilongjiang
  - Novo Nordisk Investigational Site, Chenzhou, Hunan
  - Novo Nordisk Investigational Site, Changzhou, Jiangsu
  - Novo Nordisk Investigational Site, Nanjing, Jiangsu
  - Novo Nordisk Investigational Site, Suzhou, Jiangsu
  - Novo Nordisk Investigational Site, Zhenjiang, Jiangsu
  - Novo Nordisk Investigational Site, Nanchang, Jiangxi
  - Novo Nordisk Investigational Site, Changchun, Jilin
  - Novo Nordisk Investigational Site, Yanji, Jilin
  - Novo Nordisk Investigational Site, Shenyang, Liaoning
  - Novo Nordisk Investigational Site, Yinchuan, Ningxia
  - Novo Nordisk Investigational Site, Xi'an, Shaanxi
  - Novo Nordisk Investigational Site, Jinan, Shandong
  - Novo Nordisk Investigational Site, Qingdao, Shandong
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Taiyuan, Shanxi
  - Novo Nordisk Investigational Site, Tianjin, Tianjin Municipality
  - Novo Nordisk Investigational Site, Kunming, Yunnan
  - Novo Nordisk Investigational Site, Beijing
  - Novo Nordisk Investigational Site, Changsha
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong
- South Africa (4):
  - Novo Nordisk Investigational Site, Boksburg, Gauteng
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
- South Korea (6):
  - Novo Nordisk Investigational Site, Daejeon
  - Novo Nordisk Investigational Site, Seongnam-si, Gyeonggi-do
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Suwon
  - Novo Nordisk Investigational Site, Suwon-si, Gyeonggi-do
  - Novo Nordisk Investigational Site, Wŏnju
- Taiwan (2):
  - Novo Nordisk Investigational Site, Taipei
  - Novo Nordisk Investigational Site, Taoyuan
- Ukraine (3):
  - Novo Nordisk Investigational Site, Dnipro
  - Novo Nordisk Investigational Site, Kyiv
  - Novo Nordisk Investigational Site, Lviv

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Ji L, Dong X, Li Y, Li Y, Lim S, Liu M, Ning Z, Rasmussen S, Skjoth TV, Yuan G, Eliaschewitz FG. Efficacy and safety of once-weekly semaglutide versus once-daily sitagliptin as add-on to metformin in patients with type 2 diabetes in SUSTAIN China: A 30-week, double-blind, phase 3a, randomized trial. Diabetes Obes Metab. 2021 Feb;23(2):404-414. doi: 10.1111/dom.14232. Epub 2021 Jan 3. PMID 33074557
- [Derived] Lee BW, Cho YM, Kim SG, Ko SH, Lim S, Dahaoui A, Jeong JS, Lim HJ, Yu JM. Efficacy and Safety of Once-Weekly Semaglutide Versus Once-Daily Sitagliptin as Metformin Add-on in a Korean Population with Type 2 Diabetes. Diabetes Ther. 2024 Feb;15(2):547-563. doi: 10.1007/s13300-023-01515-0. Epub 2024 Jan 18. PMID 38236431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 65 sites in 5 countries/regions as follows:
  Region China: 42 sites; Brazil: 3 sites; Republic of Korea: 12 sites; South Africa: 5 sites; Ukraine: 3 sites.
Groups:
- Semaglutide 0.5 mg: Participants took subcutaneous (s.c., under the skin) injection of semaglutide, once weekly for 30 weeks: 0.25 mg for 0-4 weeks followed by 0.5 mg for 5-30 weeks. Participants also took sitagliptin placebo (0 mg) tablet orally, once daily for 30 weeks. Both semaglutide and sitagliptin placebo were taken any time of the day irrespective of meals. Participants continued taking their pre-trial metformin with the same dose and frequency throughout the trial.
- Semaglutide 1.0 mg: Participants took subcutaneous (s.c., under the skin) injection of semaglutide, once weekly for 30 weeks: 0.25 mg for 0-4 weeks followed by 0.5 mg for 5-8 weeks and then 1.0 mg for 9-30 weeks. Participants also took sitagliptin placebo (0 mg) tablet orally, once daily for 30 weeks. Both semaglutide and sitagliptin placebo were taken any time of the day irrespective of meals. Participants continued taking their pre-trial metformin with the same dose and frequency throughout the trial.
- Sitagliptin: Participants were randomised to 2 different groups (Group 1: sitagliptin + semaglutide placebo 0.5 mg and Group 2: sitagliptin + semaglutide placebo 1.0 mg). Both groups were pooled together for data analysis. Participants took 100 mg sitagliptin tablets once-daily for 30 weeks. Participants also took semaglutide placebo injection with volume matched to different doses (0.25 mg/0.5 mg/1.0 mg) of semaglutide injection for 30 weeks. Both sitagliptin and semaglutide placebo were taken any time of the day irrespective of meals. Participants continued taking their pre-trial metformin with the same dose and frequency throughout the trial.
Period: Overall Study
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Started | 288 | 290 | 290
Exposed | 287 | 290 | 290
Full Analysis Set (FAS) | 288 | 290 | 290
Safety Analysis Set (SAS) | 287 | 290 | 290
Completed | 263 | 262 | 280
Not Completed | 25 | 28 | 10
Not completed — Withdrawal by Subject | 21 | 26 | 9
Not completed — Lost to Follow-up | 3 | 1 | 1
Not completed — Death | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set comprised of all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin | Total
Number analyzed (Participants) | 288 | 290 | 290 | 868
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.0 (11.4) | 53.0 (10.6) | 53.1 (10.4) | 53.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 136 | 105 | 369
  Male | 160 | 154 | 185 | 499
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 28 | 30 | 82
  Not Hispanic or Latino | 264 | 262 | 260 | 786
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 243 | 251 | 244 | 738
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 8 | 9 | 25
  White | 30 | 28 | 31 | 89
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 3 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change from baseline (week 0) to week 30 in glycosylated haemoglobin (HbA1c) was evaluated. Results are based on the 'on-treatment without rescue medication' observation period and 'in trial' observation period. 'On-treatment without rescue medication' observation period: started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first. 'In-trial' observation period: started when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature treatment discontinuation.
Time Frame: Week 0, week 30
Population: Full analysis set comprised of all randomised participants."Number Analyzed" = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 288 | 290 | 290
Percentage of glycosylated haemoglobin
  On-treatment without rescue medication obs. period: number analyzed (Participants) | 235 | 238 | 250
  On-treatment without rescue medication obs. period | -1.5 (1.1) | -1.8 (0.9) | -1.0 (0.9)
  In-trial observation period: number analyzed (Participants) | 256 | 258 | 278
  In-trial observation period | -1.5 (1.1) | -1.7 (1.0) | -0.9 (0.9)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Sitagliptin; The post-baseline responses are analysed using a mixed model for repeated measurements with treatment and region China/Other as fixed factors and baseline value as covariate, all nested within visit. Mean estimates are adjusted according to observed baseline distribution; Test type: Non-Inferiority — Non-inferiority was concluded if the upper limit of the two-sided 95% confidence interval for the estimated difference in HbA1c between semaglutide and sitagliptin was less than 0.3%; p < .0001, Mixed Models Analysis; Treatment difference = -0.85, 95% CI 2-sided [-1.00 to -0.70]
Statistical Analysis 2: Comparison: Semaglutide 0.5 mg vs Sitagliptin; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < .0001, Mixed Models Analysis; Treatment difference = -0.51, 95% CI 2-sided [-0.66 to -0.36]
Statistical Analysis 3: Comparison: Semaglutide 1.0 mg vs Sitagliptin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Superiority was concluded if the upper limit of the two-sided 95% confidence interval for the estimated difference in HbA1c between semaglutide and sitagliptin was below 0%; p < .0001, Mixed Models Analysis; Treatment difference = -0.85, 95% CI 2-sided [-1.00 to -0.70]
Statistical Analysis 4: Comparison: Semaglutide 0.5 mg vs Sitagliptin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 3]; p < .0001, Mixed Models Analysis; Treatment difference = -0.51, 95% CI 2-sided [-0.66 to -0.36]

2. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week 0) to week 30 in body weight was evaluated. Results are based on the 'on-treatment without rescue medication' observation period which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: Full analysis set comprised of all randomised participants. "Overall Number of Participants Analyzed" = participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 238 | 239 | 253
Kilogram (kg) | -3.0 (3.8) | -4.2 (3.7) | -0.4 (2.5)

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) to week 30 in FPG was evaluated. Results are based on the 'on-treatment without rescue medication' observation period which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: Full analysis set comprised of all randomised participants. "Overall Number of Participants Analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 237 | 238 | 253
Millimoles per liter (mmol/L) | -2.18 (2.5) | -2.62 (2.13) | -1.0 (1.74)

4. Secondary Outcome: Change in Self-measured Plasma Glucose (SMPG) - Mean 7-point Profile
Description: Change from baseline (week 0) to week 30 in SMPG mean 7-point profile was evaluated. SMPG was recorded at the following 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after dinner and at bedtime. Mean 7-point profile was defined as the area under the profile, calculated using the trapezoidal method, divided by the measurement time. Results are based on the 'on-treatment without rescue medication' observation period which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 236 | 238 | 251
Millimoles per liter (mmol/L) | -2.5 (2.4) | -3.3 (2.2) | -1.6 (2.0)

5. Secondary Outcome: Change in Self-measured Plasma Glucose (SMPG) - Mean Postprandial Increment Over All Meals
Description: Change from baseline (week 0) to week 30 in SMPG mean postprandial increment over all meals was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 234 | 237 | 251
Millimoles per liter (mmol/L) | -1.0 (2.2) | -1.2 (2.1) | -0.7 (2.2)

6. Secondary Outcome: Change in Fasting Insulin - Ratio to Baseline
Description: Change in fasting insulin from baseline (week 0) to week 30 is presented as ratio to baseline. Fasting insulin was measured in picomoles per liter (pmol/L). Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting insulin
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 229 | 237 | 254
Ratio of fasting insulin | 1.06 (46.6) | 1.03 (51.2) | 1.01 (41.6)

7. Secondary Outcome: Change in Fasting C-peptide - Ratio to Baseline
Description: Change in fasting C-peptide from baseline (week 0) to week 30 is presented as ratio to baseline. C-peptide was measured in nanomoles per liter (nmol/L). Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting C-peptide
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 234 | 239 | 254
Ratio of fasting C-peptide | 1.08 (30.3) | 1.05 (32.4) | 1.0 (32.2)

8. Secondary Outcome: Change in Fasting Glucagon - Ratio to Baseline
Description: Change in fasting glucagon from baseline (week 0) to week 30 is presented as ratio to baseline. Fasting glucagon was measured in picogram per mililiter (pg/mL). Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting glucagon
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 205 | 206 | 221
Ratio of fasting glucagon | 0.89 (32.4) | 0.89 (28.1) | 0.93 (25.0)

9. Secondary Outcome: Change in Fasting Proinsulin - Ratio to Baseline
Description: Change in fasting proinsulin from baseline (week 0) to week 30 is presented as ratio to baseline. Fasting proinsulin was measured in picomole per liter (pmol/L). Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting proinsulin
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 234 | 241 | 253
Ratio of fasting proinsulin | 0.68 (62.7) | 0.59 (65.3) | 0.81 (58.2)

10. Secondary Outcome: Change in Fasting Proinsulin/Insulin Ratio - Ratio to Baseline
Description: Change in fasting proinsulin/insulin ratio from baseline (week 0) to week 30 is presented as ratio to baseline. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting proinsulin/insulin
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 226 | 237 | 253
Ratio of fasting proinsulin/insulin | 0.63 (50.2) | 0.57 (52.1) | 0.80 (45.4)

11. Secondary Outcome: Change in Fasting HOMA-B (Beta-cell Function) - Ratio to Baseline
Description: Change in fasting HOMA-B (homeostasis model assessment beta-cell function) from baseline (week 0) to week 30 is presented as ratio to baseline. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting HOMA-B
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 228 | 236 | 252
Ratio of fasting HOMA-B | 1.81 (57.3) | 1.95 (59.1) | 1.25 (46.1)

12. Secondary Outcome: Change in Fasting HOMA-IR (Insulin Resistence) - Ratio to Baseline
Description: Change in fasting HOMA-IR (homeostasis model assessment insulin resistence) from baseline (week 0) to week 30 is presented as ratio to baseline. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting HOMA-IR
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 228 | 236 | 252
Ratio of fasting HOMA-IR | 0.81 (60.9) | 0.74 (63.2) | 0.90 (52.0)

13. Secondary Outcome: Change in Patient Reported Outcome Questionnaire: SF-36v2™ Score
Description: Short Form (SF)-36 is a 36-item patient-reported survey that measures patient's overall health-related quality of life (HRQoL). SF-36v2™ (acute version) questionnaire measured 8 domains of functional health & well-being and 2 component summary scores (physical component summary-PCS and mental component summary-MCS). The 0-100 scale scores (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively of the 2009 U.S. general population. Change from baseline (week 0) in the domain scores and component summary (PCS and MCS) scores were evaluated at weeks 30. A positive change score indicates an improvement since baseline. Results are based on the data from the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 246 | 249 | 257
Score on a scale
  Physical component summary (PCS) | 1.3 (5.9) | 1.1 (6.0) | 0.0 (5.8)
  Physical functioning | 0.6 (5.6) | 0.9 (7.4) | -0.3 (5.5)
  Role-physical | 1.4 (7.6) | 0.2 (6.9) | -0.0 (7.0)
  Bodily pain | 0.6 (8.4) | 0.4 (9.9) | 0.0 (9.8)
  General health | 3.3 (8.8) | 2.9 (9.4) | 2.2 (9.0)
  Mental component summary (MCS) | 1.2 (8.0) | 0.5 (8.4) | 1.5 (7.7)
  Social functioning | 1.3 (7.0) | -0.4 (7.8) | 0.8 (7.6)
  Role-emotional | 1.3 (8.5) | 0.9 (8.9) | 1.0 (8.6)
  Vitality | 1.2 (9.8) | 1.4 (10.1) | 1.1 (9.1)
  Mental health | 0.9 (8.7) | 0.4 (9.1) | 1.1 (7.9)

14. Secondary Outcome: Change in Patient Reported Outcome Questionnaire: DTSQs Score
Description: Change from baseline (week 0) in Diabetes Treatment Satisfaction Questionnaire (DTSQs) was evaluated at week 30. The DTSQs items are scored on a 7-point graded response scale ranging from 6 to 0. Higher scores indicate higher levels of treatment satisfaction for DTSQs items 3 -8. For items 1 and 2 a higher score indicates a higher patient perceived experience of high blood sugars and low blood sugars, respectively. Thus, lower scores indicate a perception of blood glucose levels being "none of the time" unacceptably high (item 1) or low (item 2). The domain score of total treatment satisfaction (total treatment satisfaction score) was computed by adding the six items scores 3-8. The score ranges 0-36. A higher treatment satisfaction score indicates a higher level of treatment satisfaction. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 246 | 249 | 257
Score on a scale
  1) Feeling of unacceptably high blood sugars | -1.4 (2.2) | -1.6 (2.2) | -1.0 (2.2)
  2) Feeling of unacceptably low blood sugars | -0.1 (1.9) | -0.3 (2.0) | -0.1 (1.7)
  3) Satisfaction with treatment | 1.1 (1.8) | 1.3 (1.7) | 0.7 (1.7)
  4) Convenience of treatment | 0.7 (1.6) | 0.7 (1.5) | 0.5 (1.8)
  5) Flexibility of current treatment | 0.7 (1.6) | 0.8 (1.4) | 0.4 (1.5)
  6) Satisfaction with understanding of diabetes | 0.9 (1.7) | 0.8 (1.5) | 0.7 (1.8)
  7) Recommending treatment to others | 0.9 (1.8) | 0.9 (1.6) | 0.7 (1.7)
  8) Satisfaction to continue with present treatment | 0.7 (1.6) | 0.7 (1.6) | 0.6 (1.6)
  Total Diabetic Treatment Satisfaction score | 4.9 (7.2) | 5.1 (6.3) | 3.7 (7.2)

15. Secondary Outcome: Change in High-sensitivity CRP - Ratio to Baseline
Description: Change in high-sensitivity C-reactive protein (CRP) from baseline (week 0) to week 30 is presented as ratio to baseline. High-sensitivity CRP was measured in mg/L. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of high-sensitivity CRP
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 238 | 240 | 252
Ratio of high-sensitivity CRP | 0.73 (121.2) | 0.64 (108.6) | 0.96 (128.2)

16. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline (week 0) to week 30 was measured. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 238 | 239 | 254
Centimeter (cm) | -2.7 (5.0) | -4.0 (4.8) | -0.7 (4.4)

17. Secondary Outcome: Change in BMI
Description: Change in body mass index (BMI) from baseline (week 0) to week 30 was measured. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 238 | 239 | 253
Kilogram per square meter (kg/m^2) | -1.1 (1.4) | -1.6 (1.4) | -0.1 (0.9)

18. Secondary Outcome: Change in Fasting Total Cholesterol - Ratio to Baseline
Description: Change in fasting total cholesterol from baseline (week 0) to week 30 is presented as ratio to baseline. Fasting total cholesterol was measured in mmol/L. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting total cholesterol
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 238 | 240 | 252
Ratio of fasting total cholesterol | 0.95 (20.2) | 0.95 (17.7) | 1.00 (16.8)

19. Secondary Outcome: Change in Fasting LDL Cholesterol - Ratio to Baseline
Description: Change in fasting low density lipoprotein (LDL) from baseline (week 0) to week 30 is presented as ratio to baseline. Fasting LDL was measured in mmol/L. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting LDL cholesterol
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 237 | 240 | 250
Ratio of fasting LDL cholesterol | 0.97 (33.2) | 0.99 (31.6) | 1.01 (26.1)

20. Secondary Outcome: Change in Fasting VLDL Cholesterol - Ratio to Baseline
Description: Change in fasting very low density lipoprotein (VLDL) from baseline (week 0) to week 30 is presented as ratio to baseline. Fasting VLDL was measured in mmol/L. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting VLDL cholesterol
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 237 | 240 | 251
Ratio of fasting VLDL cholesterol | 0.86 (44.8) | 0.82 (38.8) | 0.93 (46.3)

21. Secondary Outcome: Change in Fasting HDL Cholesterol - Ratio to Baseline
Description: Change in fasting high density lipoprotein (HDL) from baseline (week 0) to week 30 is presented as ratio to baseline. Fasting HDL was measured in mmol/L. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting HDL cholesterol
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 238 | 240 | 251
Ratio of fasting HDL cholesterol | 1.00 (15.8) | 1.02 (16.3) | 1.01 (14.1)

22. Secondary Outcome: Change in Fasting Triglycerides - Ratio to Baseline
Description: Change in fasting triglycerides from baseline (week 0) to week 30 is presented as ratio to baseline. Triglycerides was measured in mmol/L. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting triglycerides
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 237 | 240 | 251
Ratio of fasting triglycerides | 0.86 (47.5) | 0.81 (41.9) | 0.93 (49.1)

23. Secondary Outcome: Change in Free Fatty Acids - Ratio to Baseline
Description: Change in free fatty acids from baseline (week 0) to week 30 is presented as ratio to baseline. Free fatty acids was measured in mmol/L. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of free fatty acids
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 231 | 238 | 254
Ratio of free fatty acids | 0.78 (70.4) | 0.78 (65.8) | 0.87 (61.8)

24. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic Blood Pressure)
Description: Change from baseline (week 0) to week 30 in systolic blood pressure and diastolic blood pressure were evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 238 | 239 | 254
Millimeters of mercury (mmHg)
  Systolic blood pressure | -3.4 (14.7) | -6.5 (13.4) | -0.9 (13.6)
  Diastolic blood pressure | -0.7 (9.4) | -1.5 (8.7) | -0.8 (8.5)

25. Secondary Outcome: Percentage of Participants Who Achieved HbA1c <7.0% (53 mmol/Mol), ADA Target, (Yes/no)
Description: Percentage of participants who achieved HbA1c < 7.0% (53 millimoles per mole [mmol/mol]), American Diabetes Association (ADA) target (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 30
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 235 | 238 | 250
Percentage of participants
  Yes | 74.5 | 84.0 | 49.6
  No | 25.5 | 16.0 | 50.4

26. Secondary Outcome: Percentage of Participants Who Achieved HbA1c ≤6.5% (48 mmol/Mol), AACE Target, (Yes/no)
Description: Percentage of participants who achieved HbA1c ≤6.5% (48 millimoles per mole [mmol/mol]), American Association of Clinical Endocrinologists (AACE) target (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 30
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 235 | 238 | 250
Percentage of participants
  Yes | 60.4 | 70.6 | 31.6
  No | 39.6 | 29.4 | 68.4

27. Secondary Outcome: Percentage of Participants That Achieved (Yes/no): HbA1c <7.0% (53 mmol/Mol) Without Severe or Blood Glucose (BG)-Confirmed Symptomatic Hypoglycaemia and no Weight Gain
Description: Severe or blood glucose (BG)-confirmed symptomatic hypoglycaemia is an episode that is severe according to the American Diabetes Association classification or blood glucose-confirmed by a plasma glucose value <3.1 mmol/L (56 milligrams per deciliter [mg/dL]) with symptoms consistent with hypoglycaemia. Percentage of participants who achieved HbA1c below 7.0% (53 mmol/mol) without severe or blood glucose confirmed symptomatic hypoglycaemia episodes and no weight gain (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 30
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 235 | 238 | 249
Percentage of participants
  Yes | 66.0 | 76.9 | 33.7
  No | 34.0 | 23.1 | 66.3

28. Secondary Outcome: Percentage of Participants That Achieved (Yes/no): Body Weight Loss ≥5%
Description: Percentage of participants losing ≥5% of baseline body weight (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 30
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 238 | 239 | 253
Percentage of participants
  Yes | 36.6 | 52.7 | 5.9
  No | 63.4 | 47.3 | 94.1

29. Secondary Outcome: Percentage of Participants That Achieved (Yes/no): Body Weight Loss ≥10%
Description: Percentage of participants losing ≥10% of baseline body weight (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 30
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 238 | 239 | 253
Percentage of participants
  Yes | 9.7 | 17.2 | 0.4
  No | 90.3 | 82.8 | 99.6

30. Secondary Outcome: Total Number of Treatment Emergent Adverse Events
Description: A treatment emergent adverse event (TEAE) is defined as an adverse event with onset in the on-treatment observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0 to week 30
Population: Safety analysis set comprised of all randomised participants exposed to at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 287 | 290 | 290
Events | 729 | 788 | 596

31. Secondary Outcome: Number of Treatment Emergent Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes
Description: Hypoglycaemic episodes are defined as treatment-emergent if the onset of the episode occurs within the on-treatment observation period. Severe or BG-confirmed symptomatic hypoglycaemia is an episode that is severe according to the American Diabetes Association classification or blood glucose-confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0 to week 30
Population: Safety analysis set comprised of all randomised participants exposed to at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 287 | 290 | 290
Episodes | 3 | 7 | 5

32. Secondary Outcome: Participants With Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes
Description: Number of participants with treatment emergent severe or blood glucose-confirmed symptomatic hypoglycaemic episodes. Hypoglycaemic episodes defined as treatment-emergent if the onset of the episode occurs within the on-treatment observation period. Severe or BG-confirmed symptomatic hypoglycaemia is an episode that is severe according to the American Diabetes Association classification or blood glucose-confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0 to week 30
Population: Safety analysis set comprised of all randomised participants exposed to at least one dose of trial product.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 287 | 290 | 290
Participants | 2 | 6 | 4

33. Secondary Outcome: Change in Haematological Parameter: Haemoglobin - Ratio to Baseline
Description: Change in haemoglobin from baseline (week 0) to week 30 is presented as ratio to baseline. Haemoglobin was measured in mmol/L. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: Safety analysis set comprised of all randomised participants exposed to at least one dose of trial product. "Overall Number of Participants Analyzed" = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of haemoglobin
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 239 | 235 | 266
Ratio of haemoglobin | 1.00 (6.0) | 1.00 (5.6) | 1.00 (5.4)

34. Secondary Outcome: Change in Haematological Parameter: Haematocrit - Ratio to Baseline
Description: Change in haematocrit from baseline (week 0) to week 30 is presented as ratio to baseline. Haematocrit was measured in percentage. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of haematocrit
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 239 | 235 | 266
Ratio of haematocrit | 1.00 (6.3) | 1.00 (6.3) | 1.00 (6.3)

35. Secondary Outcome: Change in Hematological Parameter: Thrombocytes - Ratio to Baseline
Description: Change in thrombocytes from baseline (week 0) to week 30 is presented as ratio to baseline. Thrombocytes was measured in 10^9 cells per liter. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of thrombocytes
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 238 | 233 | 266
Ratio of thrombocytes | 1.01 (21.3) | 1.01 (21.2) | 0.99 (17.9)

36. Secondary Outcome: Change in Hematological Parameter: Erythrocytes - Ratio to Baseline
Description: Change in erythrocytes from baseline (week 0) to week 30 is presented as ratio to baseline. Erythrocytes were measured in 10^12 cells per liter. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of erythrocytes
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 239 | 235 | 266
Ratio of erythrocytes | 0.99 (5.6) | 0.99 (5.4) | 0.99 (5.0)

37. Secondary Outcome: Change in Hematological Parameter: Leukocytes - Ratio to Baseline
Description: Change in leukocytes from baseline (week 0) to week 30 is presented as ratio to baseline. Leukocytes were measured in 10^9 cells per liter. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of leukocytes
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 239 | 235 | 266
Ratio of leukocytes | 1.03 (21.1) | 1.01 (23.7) | 1.08 (24.9)

38. Secondary Outcome: Change in Hematological Parameter (Differential Cell Count of Leukocytes): Basophils - Ratio to Baseline
Description: Change in basophils from baseline (week 0) to week 30 is presented as ratio to baseline. Basophils were measured in percentage. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of basophils
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 229 | 230 | 251
Ratio of basophils | 0.91 (68.1) | 0.80 (71.3) | 0.83 (69.6)

39. Secondary Outcome: Change in Hematological Parameter (Differential Cell Count of Leukocytes): Neutrophils - Ratio to Baseline
Description: Change in neutrophils from baseline (week 0) to week 30 is presented as ratio to baseline. Neutrophils were measured in percentage. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of neutrophils
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 239 | 235 | 266
Ratio of neutrophils | 1.01 (12.9) | 1.02 (20.2) | 1.02 (13.7)

40. Secondary Outcome: Change in Hematological Parameter (Differential Cell Count of Leukocytes): Eosinophils - Ratio to Baseline
Description: Change in eosinophils from baseline (week 0) to week 30 is presented as ratio to baseline. Eosinophils were measured in percentage. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of eosinophils
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 238 | 234 | 265
Ratio of eosinophils | 0.98 (57.9) | 1.04 (64.7) | 1.00 (65.9)

41. Secondary Outcome: Change in Hematological Parameter (Differential Cell Count of Leukocytes): Monocytes - Ratio to Baseline
Description: Change in monocytes from baseline (week 0) to week 30 is presented as ratio to baseline. Monocytes were measured in percentage. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of monocytes
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 239 | 235 | 266
Ratio of monocytes | 0.96 (33.7) | 0.98 (34.7) | 1.04 (36.1)

42. Secondary Outcome: Change in Hematological Parameter (Differential Cell Count of Leukocytes): Lymphocytes - Ratio to Baseline
Description: Change in lymphocytes from baseline (week 0) to week 30 is presented as ratio to baseline. Lymphocytes were measured in percentage. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lymphocytes
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 239 | 235 | 266
Ratio of lymphocytes | 1.01 (22.7) | 0.98 (23.6) | 0.97 (24.2)

43. Secondary Outcome: Change in Biochemistry Parameter: Amylase - Ratio to Baseline
Description: Change in amylase from baseline (week 0) to week 30 is presented as ratio to baseline. Amylase was measured in units per liter (U/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 247 | 242 | 271
Ratio of amylase | 1.17 (30.6) | 1.19 (23.6) | 1.10 (22.5)

44. Secondary Outcome: Change in Biochemistry Parameter: Lipase - Ratio to Baseline
Description: Change in lipase from baseline (week 0) to week 30 is presented as ratio to baseline. Lipase was measured in units per liter (U/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 247 | 243 | 273
Ratio of lipase | 1.33 (43.9) | 1.42 (51.2) | 1.24 (47.2)

45. Secondary Outcome: Change in Biochemistry Parameter: Alkaline Phosphatase - Ratio to Baseline
Description: Change in alkaline phosphatase from baseline (week 0) to week 30 is presented as ratio to baseline. Alkaline phosphatase was measured in units per liter (U/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of alkaline phosphatase
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 247 | 242 | 271
Ratio of alkaline phosphatase | 0.92 (31.3) | 0.91 (15.3) | 0.92 (20.1)

46. Secondary Outcome: Change in Biochemistry Parameter: Alanine Aminotransferase - Ratio to Baseline
Description: Change in alanine aminotransferase from baseline (week 0) to week 30 is presented as ratio to baseline. Alanine aminotransferase was measured in units per liter (U/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of alanine aminotransferase
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 246 | 241 | 269
Ratio of alanine aminotransferase | 0.86 (55.7) | 0.83 (47.1) | 0.95 (35.1)

47. Secondary Outcome: Change in Biochemistry Parameter: Aspartate Aminotransferase - Ratio to Baseline
Description: Change in aspartate aminotransferase from baseline (week 0) to week 30 is presented as ratio to baseline. Aspartate aminotransferase was measured in units per liter (U/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: Safety analysis set comprised of all randomised participants exposed to at least one dose of trial product. "Overall Number of Participants Analyzed "= participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of aspartate aminotransferase
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 246 | 242 | 268
Ratio of aspartate aminotransferase | 0.92 (36.9) | 0.88 (36.7) | 0.99 (29.3)

48. Secondary Outcome: Change in Biochemistry Parameter: Total Bilirubin - Ratio to Baseline
Description: Change in total bilirubin from baseline (week 0) to week 30 is presented as ratio to baseline. Total bilirubin was measured in micromoles per liter (umol/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total bilirubin
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 247 | 241 | 269
Ratio of total bilirubin | 0.93 (32.8) | 0.93 (35.4) | 0.93 (36.4)

49. Secondary Outcome: Change in Biochemistry Parameter: Calcium (Corrected)- Ratio to Baseline
Description: Change in calcium (corrected) from baseline (week 0) to week 30 is presented as ratio to baseline. Calcium was measured in millimoles per litre (mmol/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcium
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 247 | 242 | 271
Ratio of calcium | 1.01 (3.7) | 1.01 (3.2) | 1.01 (3.4)

50. Secondary Outcome: Change in Biochemistry Parameter: Total Calcium - Ratio to Baseline
Description: Change in total calcium from baseline (week 0) to week 30 is presented as ratio to baseline. Calcium was measured in millimoles per litre (mmol/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total calcium
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 247 | 242 | 271
Ratio of total calcium | 1.02 (4.4) | 1.01 (3.8) | 1.01 (3.9)

51. Secondary Outcome: Change in Biochemistry Parameter: Potassium - Ratio to Baseline
Description: Change in potassium from baseline (week 0) to week 30 is presented as ratio to baseline. Potassium was measured in millimoles per liter (mmol/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of potassium
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 246 | 242 | 271
Ratio of potassium | 1.01 (7.7) | 1.00 (8.4) | 1.00 (8.5)

52. Secondary Outcome: Change in Biochemistry Parameter: Sodium - Ratio to Baseline
Description: Change in sodium from baseline (week 0) to week 30 is presented as ratio to baseline. Sodium was measured in millimoles per litre (mmol/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of sodium
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 246 | 242 | 271
Ratio of sodium | 1.01 (1.5) | 1.00 (1.5) | 1.00 (1.4)

53. Secondary Outcome: Change in Biochemistry Parameter: Albumin - Ratio to Baseline
Description: Change in albumin from baseline (week 0) to week 30 is presented as ratio to baseline. Albumin was measured in grams per deciliter (g/dL). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of albumin
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 247 | 242 | 271
Ratio of albumin | 1.02 (5.4) | 1.02 (5.4) | 1.01 (4.8)

54. Secondary Outcome: Change in Biochemistry Parameter: Creatine Kinase - Ratio to Baseline
Description: Change in creatine kinase from baseline (week 0) to week 30 is presented as ratio to baseline. Creatine kinase was measured in units per liter (U/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of creatine kinase
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 247 | 242 | 270
Ratio of creatine kinase | 1.02 (49.1) | 0.96 (41.8) | 1.07 (43.5)

55. Secondary Outcome: Change in Biochemistry Parameter: Total Protein- Ratio to Baseline
Description: Change in Total protein from baseline (week 0) to week 30 is presented as ratio to baseline. Total Protein was measured in grams per deciliter (g/dL). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total protein
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 247 | 242 | 271
Ratio of total protein | 1.01 (5.0) | 1.00 (5.3) | 1.01 (5.2)

56. Secondary Outcome: Change in Biochemistry Parameter: Creatinine - Ratio to Baseline
Description: Change in creatinine from baseline (week -2) to week 30 is presented as ratio to baseline. Creatinine was measured in micromoles per lier (umol/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week -2, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of creatinine
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 247 | 243 | 273
Ratio of creatinine | 1.08 (12.6) | 1.07 (11.7) | 1.05 (12.1)

57. Secondary Outcome: Change in Biochemistry Parameter: Urea - Ratio to Baseline
Description: Change in urea from baseline (week 0) to week 30 is presented as ratio to baseline. Urea was measured in millimoles per liter (mmol/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of urea
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 247 | 243 | 273
Ratio of urea | 1.01 (25.6) | 1.02 (26.4) | 1.01 (23.6)

58. Secondary Outcome: Change in Biochemistry Parameter: Estimated Glomerular Filtration Rate (eGFR) - Ratio to Baseline
Description: Change in estimated glomerular filtration rate (eGFR) from baseline (week 0) to week 30 is presented as ratio to baseline. Glomerular filtration rate was measured in milliliter/minute/specific surface area (mL/min/SSA). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of eGFR
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 247 | 243 | 273
Ratio of eGFR | 0.92 (14.6) | 0.92 (13.6) | 0.94 (14.0)

59. Secondary Outcome: Change in Calcitonin - Ratio to Baseline
Description: Change in calcitonin from baseline (week -2) to week 30 is presented as ratio to baseline. Calcitonin was measured in nanogram per liter (ng/L). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week -2, week 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcitonin
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 246 | 244 | 273
Ratio of calcitonin | 0.96 (37.5) | 1.00 (44.8) | 0.96 (48.4)

60. Secondary Outcome: Change in Urinalysis Parameter - UACR-ratio to Baseline
Description: Change in urin albumin to creatinine ratio (UACR) from baseline (week 0) to week 30 is presented as ratio to baseline. UACR was measured in milligram/millimole (mg/mmol). Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: Safety analysis set comprised of all randomised participants exposed to at least one dose of trial product. "Overall Number of Participants Analyzed"=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of UACR
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 155 | 164 | 189
Ratio of UACR | 0.77 (83.5) | 0.69 (78.4) | 0.89 (76.0)

61. Secondary Outcome: Change in Urinalysis Parameter: Glucose
Description: Glucose in urine was assessed by the investigator and categorised as negative, [100-249], [250-499], [500-999] and >= 1000. Number of participants in each category at baseline (week 0) and week 30 are presented. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 286 | 289 | 287
Participants
  At week 0: Negative | 189 | 187 | 176
  At week 0: 100-249 | 28 | 27 | 42
  At week 0: 250-499 | 12 | 20 | 25
  At week 0: 500-999 | 20 | 25 | 21
  At week 0: >= 1000 | 37 | 30 | 23
  At week 30: Negative | 244 | 258 | 233
  At week 30: 100-249 | 7 | 15 | 23
  At week 30: 250-499 | 10 | 5 | 5
  At week 30: 500-999 | 11 | 4 | 12
  At week 30: >= 1000 | 14 | 7 | 14

62. Secondary Outcome: Change in Urinalysis Parameter: pH
Description: pH in urine was assessed by the investigator and categorised as 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, >=9. Number of participants in each category at baseline (week 0) and week 30 are presented. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 286 | 289 | 287
Participants
  At week 0: 5 | 0 | 0 | 0
  At week 0: 5.5 | 17 | 15 | 14
  At week 0: 6 | 220 | 214 | 222
  At week 0: 6.5 | 31 | 40 | 33
  At week 0: 7 | 13 | 14 | 15
  At week 0: 7.5 | 3 | 4 | 1
  At week 0: 8 | 0 | 2 | 1
  At week 0: 8.5 | 1 | 0 | 1
  At week 0: >= 9 | 1 | 0 | 0
  At week 30: 5 | 0 | 0 | 0
  At week 30: 5.5 | 16 | 21 | 30
  At week 30: 6 | 209 | 194 | 201
  At week 30: 6.5 | 33 | 40 | 24
  At week 30: 7 | 24 | 30 | 22
  At week 30: 7.5 | 2 | 3 | 5
  At week 30: 8 | 1 | 1 | 5
  At week 30: 8.5 | 1 | 0 | 0
  At week 30: >= 9 | 0 | 0 | 0

63. Secondary Outcome: Change in Urinalysis Parameter: Protein
Description: Protein in urine was assessed by the investigator and categorised as negative, trace, 30-99, 100-299, Approximately 300, >=300. Number of participants in each category at baseline (week 0) and week 30 are presented. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 286 | 289 | 287
Participants
  At week 0: Negative | 231 | 233 | 235
  At week 0: Trace | 31 | 32 | 30
  At week 0: 30-99 | 17 | 18 | 15
  At week 0: 100-299 | 6 | 4 | 6
  At week 0: Approximately 300 | 0 | 0 | 0
  At week 0: >=300 | 1 | 2 | 1
  At week 30: Negative | 247 | 248 | 239
  At week 30: Trace | 22 | 28 | 24
  At week 30: 30-99 | 13 | 9 | 12
  At week 30: 100-299 | 4 | 4 | 11
  At week 30: Approximately 300 | 0 | 0 | 0
  At week 30: >=300 | 0 | 0 | 1

64. Secondary Outcome: Change in Urinalysis Parameter: Ketones
Description: Ketones in urine was assessed by the investigator and categorised as negative, trace, 15-39, 40-79, Approximately 80, >= 80. Number of participants in each category at baseline (week 0) and week 30 are presented. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 286 | 289 | 287
Participants
  At week 0: Negative | 267 | 268 | 274
  At week 0: Trace | 11 | 17 | 9
  At week 0: 15-39 | 8 | 3 | 3
  At week 0: 40- 79 | 0 | 1 | 0
  At week 0: Approximately 80 | 0 | 0 | 1
  At week 0: >=80 | 0 | 0 | 0
  At week 30: Negative | 268 | 274 | 274
  At week 30: Trace | 12 | 12 | 11
  At week 30: 15-39 | 6 | 3 | 1
  At week 30: 40- 79 | 0 | 0 | 1
  At week 30: Approximately 80 | 0 | 0 | 0
  At week 30: >=80 | 0 | 0 | 0

65. Secondary Outcome: Change in Urinalysis Parameter: Erythrocytes
Description: Erythrocytes in urine was assessed by the investigator and categorised as negative, trace, small, moderate, large. Number of participants in each category at baseline (week 0) and week 30 are presented. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 286 | 289 | 287
Participants
  At week 0: Negative | 251 | 250 | 253
  At week 0: Trace | 25 | 20 | 19
  At week 0: Small | 5 | 8 | 9
  At week 0: Moderate | 1 | 3 | 3
  At week 0: Large | 4 | 8 | 3
  At week 30: Negative | 258 | 259 | 252
  At week 30: Trace | 18 | 13 | 22
  At week 30: Small | 4 | 5 | 9
  At week 30: Moderate | 2 | 6 | 1
  At week 30: Large | 4 | 6 | 3

66. Secondary Outcome: Change in Clinical Evaluation: Pulse
Description: Change in pulse from baseline (week 0) to week 30 is presented. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 60
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 247 | 243 | 273
Beats per minute (beats/min) | 3.7 (10.1) | 3.7 (9.4) | 0.2 (9.0)

67. Secondary Outcome: Change in Clinical Evaluation: ECG
Description: The electrocardiogram (ECG) was assessed by the investigator and categorised as normal, abnormal not clinically significant (NCS) or abnormal clinically significant (CS). Number of participants in each ECG category at baseline and week 30 are presented. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: Safety analysis set comprised of all randomised participants exposed to at least one dose of trial product. "Number Analyzed" = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 286 | 290 | 290
Participants
  At week 0: Normal | 191 | 196 | 185
  At week 0: Abnormal, NCS | 72 | 68 | 76
  At week 0: Abnormal, CS | 23 | 26 | 29
  At week 30: number analyzed (Participants) | 262 | 264 | 278
  At week 30: Normal | 162 | 172 | 167
  At week 30: Abnormal, NCS | 81 | 74 | 85
  At week 30: Abnormal, CS | 19 | 18 | 26

68. Secondary Outcome: Change in Clinical Evaluation: Eye Examinations
Description: Eye examination was performed by the investigator and the results of the examination were interpreted for each eye (left/right) are categorised as normal, abnormal not clinically significant (NCS) or abnormal clinically significant (CS). Number of participants in each category at baseline (week 0) and at week 30 are presented. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 30
Population: as for outcome 67
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 286 | 290 | 290
Participants
  At week 0, Left eye: Normal | 202 | 222 | 202
  At week 0, Left eye: Abnormal, NCS | 40 | 32 | 47
  At week 0, Left eye: Abnormal, CS | 44 | 36 | 41
  At week 30, Left eye: number analyzed (Participants) | 230 | 233 | 247
  At week 30, Left eye: Normal | 162 | 184 | 174
  At week 30, Left eye: Abnormal, NCS | 26 | 18 | 32
  At week 30, Left eye: Abnormal, CS | 42 | 31 | 41
  At week 0, Right eye: Normal | 210 | 222 | 201
  At week 0, Right eye: Abnormal, NCS | 37 | 31 | 47
  At week 0, Right eye: Abnormal, CS | 39 | 37 | 42
  At week 52, Right eye: number analyzed (Participants) | 230 | 233 | 246
  At week 52, Right eye: Normal | 161 | 180 | 172
  At week 52, Right eye: Abnormal, NCS | 27 | 19 | 31
  At week 52, Right eye: Abnormal, CS | 42 | 34 | 43

69. Secondary Outcome: Change in Physical Examination
Description: Physical examination parameters are categorised as general appearance; nervous system (central and peripheral); cardiovascular system; gastrointestinal system; skin; respiratory system; lymph node palpation; thyroid gland; left foot; right foot; left leg and right leg. The number of participants assessed as normal, abnormal not clinically significant (NCS) and abnormal clinically significant (CS) at baseline (week -2) and week 30 are presented. Results are based on the 'on-treatment' observation period. On-treatment observation period is defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week -2, week 30
Population: as for outcome 67
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 287 | 290 | 290
Participants
  At week -2, General Appearance: Normal | 282 | 283 | 281
  At week -2, General Appearance: Abnormal, NCS | 3 | 7 | 8
  At week -2, General Appearance: Abnormal, CS | 2 | 0 | 1
  At week 30, General Appearance: number analyzed (Participants) | 256 | 253 | 276
  At week 30, General Appearance: Normal | 252 | 250 | 270
  At week 30, General Appearance: Abnormal, NCS | 3 | 3 | 5
  At week 30, General Appearance: Abnormal, CS | 1 | 0 | 1
  At week -2, Nervous System: Normal | 277 | 287 | 279
  At week -2, Nervous System: Abnormal, NCS | 5 | 1 | 8
  At week -2, Nervous System: Abnormal, CS | 5 | 2 | 3
  At week 30, Nervous System: number analyzed (Participants) | 256 | 253 | 276
  At week 30, Nervous System: Normal | 247 | 250 | 268
  At week 30, Nervous System: Abnormal, NCS | 4 | 1 | 5
  At week 30, Nervous System: Abnormal, CS | 5 | 2 | 3
  At week -2, Cardiovascular System: Normal | 276 | 281 | 278
  At week -2, Cardiovascular System: Abnormal, NCS | 9 | 6 | 10
  At week -2, Cardiovascular System: Abnormal, CS | 2 | 3 | 2
  At week 30, Cardiovascular System: number analyzed (Participants) | 256 | 253 | 276
  At week 30, Cardiovascular System: Normal | 245 | 246 | 265
  At week 30, Cardiovascular System: Abnormal, NCS | 8 | 4 | 10
  At week 30, Cardiovascular System: Abnormal, CS | 3 | 3 | 1
  At week -2, Gastrointestinal System: Normal | 280 | 285 | 280
  At week -2, Gastrointestinal System: Abnormal, NCS | 6 | 5 | 10
  At week -2, Gastrointestinal System: Abnormal, CS | 1 | 0 | 0
  At week 30, Gastrointestinal System: number analyzed (Participants) | 256 | 253 | 276
  At week 30, Gastrointestinal System: Normal | 251 | 250 | 264
  At week 30, Gastrointestinal System: Abnormal, NCS | 5 | 2 | 11
  At week 30, Gastrointestinal System: Abnormal, CS | 0 | 1 | 1
  At week -2, Musculoskeletal System: Normal | 281 | 283 | 282
  At week -2, Musculoskeletal System: Abnormal, NCS | 6 | 5 | 6
  At week -2, Musculoskeletal System: Abnormal, CS | 0 | 2 | 2
  At week 30, Musculoskeletal System: number analyzed (Participants) | 256 | 253 | 276
  At week 30, Musculoskeletal System: Normal | 252 | 247 | 270
  At week 30, Musculoskeletal System: Abnormal, NCS | 3 | 4 | 3
  At week 30, Musculoskeletal System: Abnormal, CS | 1 | 2 | 3
  At week -2, Skin: Normal | 253 | 252 | 254
  At week -2, Skin: Abnormal, NCS | 28 | 37 | 29
  At week -2, Skin: Abnormal, CS | 6 | 1 | 7
  At week 30, Skin: number analyzed (Participants) | 256 | 253 | 276
  At week 30, Skin: Normal | 226 | 217 | 240
  At week 30, Skin: Abnormal, NCS | 25 | 33 | 31
  At week 30, Skin: Abnormal, CS | 5 | 3 | 5
  At week -2, Head,Ears,Eyes,Nose, Throat, Neck: Normal | 273 | 281 | 277
  At week -2, Head,Ears,Eyes,Nose, Throat, Neck: Abnormal, NCS | 12 | 7 | 7
  At week -2, Head,Ears,Eyes,Nose, Throat, Neck: Abnormal, CS | 2 | 2 | 6
  At week 30, Head,Ears,Eyes,Nose, Throat, Neck: number analyzed (Participants) | 256 | 253 | 276
  At week 30, Head,Ears,Eyes,Nose, Throat, Neck: Normal | 245 | 244 | 263
  At week 30, Head,Ears,Eyes,Nose, Throat, Neck: Abnormal, NCS | 9 | 7 | 8
  At week 30, Head,Ears,Eyes,Nose, Throat, Neck: Abnormal, CS | 2 | 2 | 5
  At week -2, Respiratory System: Normal | 287 | 288 | 287
  At week -2, Respiratory System: Abnormal, NCS | 0 | 1 | 2
  At week -2, Respiratory System: Abnormal, CS | 0 | 1 | 1
  At week 30, Respiratory System: number analyzed (Participants) | 256 | 253 | 276
  At week 30, Respiratory System: Normal | 255 | 250 | 274
  At week 30, Respiratory System: Abnormal, NCS | 1 | 2 | 2
  At week 30, Respiratory System: Abnormal, CS | 0 | 1 | 0
  At week -2, Lymph Node Palpation: Normal | 284 | 284 | 285
  At week -2, Lymph Node Palpation: Abnormal, NCS | 2 | 5 | 4
  At week -2, Lymph Node Palpation: Abnormal, CS | 1 | 1 | 1
  At week 30, Lymph Node Palpation: number analyzed (Participants) | 256 | 253 | 276
  At week 30, Lymph Node Palpation: Normal | 255 | 250 | 271
  At week 30, Lymph Node Palpation: Abnormal, NCS | 1 | 3 | 5
  At week 30, Lymph Node Palpation: Abnormal, CS | 0 | 0 | 0
  At week -2, Thyroid Gland: Normal | 280 | 285 | 281
  At week -2, Thyroid Gland: Abnormal, NCS | 6 | 3 | 9
  At week -2, Thyroid Gland: Abnormal, CS | 1 | 2 | 0
  At week 30, Thyroid Gland: number analyzed (Participants) | 256 | 253 | 276
  At week 30, Thyroid Gland: Normal | 253 | 249 | 270
  At week 30, Thyroid Gland: Abnormal, NCS | 2 | 2 | 5
  At week 30, Thyroid Gland: Abnormal, CS | 1 | 2 | 1

70. Secondary Outcome: Anti-semaglutide Antibody Levels
Description: This outcome measure is only applicable for the semaglutide arms. Anti-semaglutide antibody level at week 30 and week 35 are presented. Antibody levels were measured in percentage of bound radioactivity-labelled semaglutide/total added radioactivity-labelled semaglutide (%B/T; B =Bound, T = Total). Evaluation was based on 'in trial' observation period, which is the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature treatment discontinuation.
Time Frame: week 30, week 35
Population: as for outcome 60
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg
Number analyzed (Participants) | 0 | 3
%B/T
  At week 30: number analyzed (Participants) | 0 | 2
  At week 30 |  | 2.8 (0.2)
  At week 35 |  | 3.3 (0.7)

71. Secondary Outcome: Occurence of Anti-semaglutide Antibodies (Yes/no)
Description: This outcome measure is only applicable for the semaglutide arms. Development of anti-semaglutide antibodies was evaluated in participants during the study. The number of participants who were positive/ negative for anti-semaglutide antibodies were presented. Evaluation was based on 'in trial' observation period, which is the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature treatment discontinuation.
Time Frame: Week 0, week 16, week 30, week 35
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg
Number analyzed (Participants) | 287 | 290
Participants
  At week 0: number analyzed (Participants) | 285 | 289
  At week 0: Yes (positive for antibody) | 0 | 1
  At week 0: No (negative for antibody) | 285 | 288
  At week 16: number analyzed (Participants) | 285 | 290
  At week 16: Yes (positive for antibody) | 1 | 0
  At week 16: No (negative for antibody) | 284 | 290
  At week 30: number analyzed (Participants) | 257 | 263
  At week 30: Yes (positive for antibody) | 0 | 2
  At week 30: No (negative for antibody) | 257 | 261
  At week 35: number analyzed (Participants) | 262 | 264
  At week 35: Yes (positive for antibody) | 0 | 3
  At week 35: No (negative for antibody) | 262 | 261

72. Secondary Outcome: Occurence of Anti-semaglutide Antibodies With In-vitro Neutralising Effect (Yes/no)
Description: This outcome measure is only applicable for the semaglutide arms. Development of anti-semaglutide antibodies with in-vitro neutralising effect was evaluated in participants during the study. The number of participants who were positive/ negative for anti-semaglutide antibodies with in vitro neutralising effect are presented. Evaluation was based on in-trial observation period, which is the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature treatment discontinuation.
Time Frame: Week 0, week 16, week 30, week 35
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg
Number analyzed (Participants) | 287 | 290
Participants
  At week 0: number analyzed (Participants) | 285 | 289
  At week 0: Yes (positive for antibody) | 0 | 0
  At week 0: No (negative for antibody) | 285 | 289
  At week 16: number analyzed (Participants) | 285 | 290
  At week 16: Yes (positive for antibody) | 0 | 0
  At week 16: No (negative for antibody) | 285 | 290
  At week 30: number analyzed (Participants) | 257 | 263
  At week 30: Yes (positive for antibody) | 0 | 0
  At week 30: No (negative for antibody) | 257 | 263
  At week 35: number analyzed (Participants) | 262 | 264
  At week 35: Yes (positive for antibody) | 0 | 0
  At week 35: No (negative for antibody) | 262 | 264

73. Secondary Outcome: Occurence of Anti-semaglutide Antibodies Cross Reacting With Endogenous GLP-1 (Yes/no)
Description: This outcome measure is only applicable for the semaglutide arms. Development of anti-semaglutide antibodies cross reacting with endogenous glucagon-like peptide-1 (GLP-1) was evaluated in participants. The number of participants who were positive/ negative for anti-semaglutide antibodies cross reacting with endogenous GLP-1 are presented. Evaluation was based on in-trial observation period, which is the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature treatment discontinuation.
Time Frame: Week 35
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg
Number analyzed (Participants) | 262 | 264
Participants
  Yes (positive for antibody) | 0 | 1
  No (negative for antibody) | 262 | 263

74. Secondary Outcome: Occurence of Cross Reacting Antibodies With in Vitro Neutralising Effect to Endogenous GLP-1 (Yes/no)
Description: This outcome measure is only applicable for the semaglutide arms. Development of cross reacting antibodies with in-vitro neutralising effect to endogenous glucagon-like peptide-1 (GLP-1) was evaluated in participants. The number of participants who were positive/ negative for anti-semaglutide antibodies with in vitro neutralising effect to endogenous GLP-1 are presented. Evaluation was based on in-trial observation period, which is the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature treatment discontinuation.
Time Frame: Week 35
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg
Number analyzed (Participants) | 262 | 264
Participants
  Yes (positive for antibody) | 0 | 0
  No (negative for antibody) | 262 | 264

ADVERSE EVENTS:
Time Frame: From the date of first dose of trial product (week 0) to end of treatment (week 30) + post treatment follow-up of 5 weeks.
Description: Evaluation of safety was based on safety analysis set (SAS) comprised of all randomised participants exposed to at least one dose of trial product.
  AEs with onset during the on-treatment observation period (the period when participants were exposed to trial product) were considered treatment-emergent.
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
All-Cause Mortality (participants affected / at risk) | 1/287 | 1/290 | 0/290
Serious Adverse Events (participants affected / at risk) | 18/287 | 19/290 | 12/290
Other Adverse Events (participants affected / at risk) | 135/287 | 139/290 | 89/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=287) | Semaglutide 1.0 mg (N=290) | Sitagliptin (N=290)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic hepatitis B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperaldosteronism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Mixed deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Neurosurgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Venous aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=287) | Semaglutide 1.0 mg (N=290) | Sitagliptin (N=290)
Abdominal discomfort (Gastrointestinal disorders) | 8 (9) | 15 (16) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 21 (21) | 23 (23) | 4 (4)
Diabetic retinopathy (Eye disorders) | 18 (18) | 14 (14) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 58 (94) | 49 (99) | 20 (24)
Lipase increased (Investigations) | 22 (30) | 13 (15) | 22 (30)
Nasopharyngitis (Infections and infestations) | 17 (21) | 9 (12) | 11 (15)
Nausea (Gastrointestinal disorders) | 22 (24) | 39 (54) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 28 (37) | 38 (45) | 43 (64)
Vomiting (Gastrointestinal disorders) | 14 (16) | 19 (22) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT03061214/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT03061214/SAP_001.pdf